CLINICAL TRIAL: NCT02730468
Title: SEP-SEQ Trial - Determining the Etiology of Sepsis Using an Infectious Disease Diagnostic Sequencing Assay
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 001-CL-01
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the performance of the Karius Infectious Diseases Plasma Sequencing Assay in patients who present to the emergency room with sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Meet 2 of 4 sepsis criteria

   1. Temperature > 38C or < 36C
   2. Heart rate > 90 bpm
   3. Respiratory rate >20 or PaCO2 <32mmHg
   4. WBC >12000/µL or < 4000/µL or > 10% bands

Exclusion Criteria:

1. Inability to understand instructions and comply with study-related procedures
2. Any condition that in the opinion of the treating physician will prevent the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be at least 18 years of age and who present to the Emergency Department with the diagnosis of sepsis
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of sequencing assay in diagnosing etiology of sepsis | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Yang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided